CLINICAL TRIAL: NCT01692665
Title: Changes of Keratometric Value and Ocular Aberration After Treatment of Meibomian Gland Dysfunction
Status: Withdrawn | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2012-0031
Record Dates: First submitted 2012-09-16; First posted 2012-09-25 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Moderate and Severe Meibomiang Gland Dysfunction (Stage 3 or Stage 4 Meibomiang Gland Dysfunction)
Keywords: meibomian gland dysfunction; keratometric value; ocular aberration
MeSH Terms: conditions — Lymphoma, Follicular; Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- stage 3 or stage 4 meibomiang gland dysfunction patients: stage 3 or stage 4 meibomiang gland dysfunction patients

SUMMARY:
Ocular aberration may play a role in determining optical quality. Recently performed study reported that ocular aberration of preocular tear film would be important factor in not only diagnosing the dry eye but also determining the efficacy of treatment. Therefore, in this study, the investigators will aim to prove the improvement of quality of vision via ocular aberration changes indirectly after the proper treatment for moderate and severe meibomian gland dysfunction. Also, the investigators will evaluate the changes of keratometric values after treatment for moderate and severe meibomian gland dysfunction, which could be demonstrated by autokeratometry, IOLMaster, Pentacam, and iTrace.

ELIGIBILITY:
Inclusion Criteria:

(1) stage 3 or 4 meibomian gland dysfunction

Exclusion Criteria:

1. history of previous ocular or intraocular surgery
2. ocular infection, non dry eye ocular inflammation, ocular allergy, autoimmune disease,
3. history of intolerance or hypersensitivity to any component of the study medications,
4. wearing contact lenses during the study period, presence of current punctal occlusion,
5. pregnancy, lactating women, and children.
6. Additionally, patients were excluded if they were using any topical ocular or systemic medication that could be used for the treatment MGD or dry eye, including topical or oral antibiotics, topical cyclosporine A, topical or oral steroids, topical non-steroidal anti-inflammatory drugs, topical ocular allergy medications or artificial tears

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stage 3 or stage 4 meibomiang gland dysfunction patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes of keratometric value and ocular aberration | a minimum of four minutes, once or twice dailybefore treatment, after 1 month, and after 2 months of treatment